CLINICAL TRIAL: NCT07023601
Title: Sentinel Node Biopsy in Relapsed Vulvar Cancer. VULCA-NODE Study.
Brief Title: International Prospective Multicentre Study That Evaluate the Sentinel Lymph Node Detection Rate in Patients With First Local Recurrent Scamous Cell Carcinoma of the Vulva.
Acronym: VULCA-NODE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Myriam Gracia, Myriam Gracia and Ignacio Zapardiel, Hospital Universitario La Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HULP: PI-6605
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Recurent Vulvar Carcinoma
MeSH Terms: interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First local recurrent vulvar carcinoma (Experimental)
  Interventions: Other: Sentinel Lymph Node Biopsy in first local recurrent vulvar carcinoma

INTERVENTIONS:
Other: Sentinel Lymph Node Biopsy in first local recurrent vulvar carcinoma — All patients will undergo a local tumor radical excision and unilateral (if medial border > 1 cm from midline) or bilateral (medial border < or equal to 1 cm from midline) Sentinel Lymph Node procedure, followed by bilateral Inguinophemoral lymphadenectomy. .

SUMMARY:
Acronym: VULCA-NODE Study Title: Sentinel Node Biopsy in Relapsed Vulvar Cancer Primary Objetive: To evaluate the SLN detection rate in the first recurrent vulvar carcinoma setting.

Secondary Objetives:

* To compare the utility of different tracers in the detection of SLN for recurrent disease and the injection pattern.
* To evaluate the surgical complications rate.
* To analyze the nodal status by ultrastaging .
* To assess the disease free and overall survival at 24 months from the first recurrence, as well as the dissemination pattern after the procedure.

Study Design: International prospective multicentre study

Inclusion Criteria:

* First local recurrent squamous cell carcinoma of the vulva (SCC).
* Unifocal, smaller or equal than 4 cm vulvar tumor not involving urethra, vagina or anus.
* No distant or groin metastasis.
* To be able to understand the study and sign informed consent.
* Over 18 years old.
* To be able to undergo planned follow up.

Exclusion Criteria:

* Multifocal recurrent disease of the vulva.
* Previous bilateral IFL.
* Synchronous, non-curable second malignancy. Timing: 4 years

ELIGIBILITY:
Inclusion Criteria:

* First local recurrent squamous cell carcinoma of the vulva (SCC).
* Unifocal, smaller or equal than 4 cm vulvar tumor not involving urethra, vagina or anus.
* No distant or groin metastasis.
* To be able to understand the study and sign informed consent.
* Over 18 years old.
* To be able to undergo planned follow up.

Exclusion Criteria:

* Multifocal recurrent disease of the vulva.
* Previous bilateral IFL.
* Synchronous, non-curable second malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the SLN detection rate in the first recurrent vulvar carcinoma setting. | From enrollment to the first 30 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided